CLINICAL TRIAL: NCT05957211
Title: Improving Drop Instillation Comfort of a Cyclosporine A Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 45135
Record Dates: First submitted 2023-06-15; First posted 2023-07-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Disease
Keywords: dry eye disease; cyclosporine; eye drop
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants will have a refrigerated 0.09% cyclosporine drop instilled in one eye, and a non-refrigerated 0.09% cyclosporine drop instilled in the other eye. The eye that receives the refrigerated drop is randomly determined.
  Interventions: Drug: 0.09% cyclosporine A ophthalmic solution

INTERVENTIONS:
Drug: 0.09% cyclosporine A ophthalmic solution — Cequa is an ophthalmic solution used to treat moderate to severe dry eye disease. The typical dosage is one drop in each eye, twice a day. The drug is packaged in sterile, single use bottles.
  Other Names: Cequa

SUMMARY:
Patients who suffer from dry eye disease are often prescribed eye drops containing cyclosporine A that help with reducing inflammation. The newest eye drop containing cyclosporine A is called Cequa (Sun Pharma, Canada). Unfortunately, nearly a quarter of (24.2%) of patients using Cequa have reported some form of discomfort (burning and stinging) when instilling the drops. This potentially discourages patients from continuing the eye drop, which prevents their dry eye disease from being managed effectively. This study is trying to determine if refrigerating the eye drops would allow the drops to feel more comfortable when they are instilled in the eye.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Ocular Surface Disease Index score >= 23.
* Strip meniscometry < 5 mm.

Exclusion Criteria:

* Contact lens wearers.
* Have corneal neuropathic or neurotrophic disease.
* Have an ocular or medical condition or taking medications that could confound a study outcome.
* Currently pregnant or breastfeeding (cyclosporine is a FDA pregnancy Category C drug).
* Have an ocular or medical condition for which Cequa is contraindicated (e.g., allergy to cyclosporine or other ingredients in Cequacurrent eye infection, cancer or precancerous condition in or around the eyes).
* Have an allergy to fluorescein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Ocular discomfort score. A subjective questionnaire that queries participants' ocular discomfort. The instrument ranges from 0 (no discomfort) to 10 (maximum discomfort). | Within 10 minutes of drop instillation
  Difference in ocular discomfort between the eye that receives a refrigerated Cequa drop and the eye that receives a non-refrigerated (room temperature) drop.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No